CLINICAL TRIAL: NCT06385522
Title: A Phase 1, First-In-Human, Open-Label, Dose-Escalating Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Ascending Intravenous Doses of BITR2101 (Anti-TNFR2) in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma Including Cutaneous and Peripheral T Cell Lymphoma
Brief Title: A Clinical Trial in Adults With Non-Hodgkin Lymphoma (NHL), With a Particular Emphasis on Cutaneous T Cell Lymphoma (CTCL), Testing the Safety and Activity of a Novel Drug to Inhibit a Protein Called Tumor Necrosis Factor Receptor 2 That Drives Both Lymphoma Growth and Escape of the Immune System
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Immune Technologies and Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BITR2101-C-01
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: NHL; Cutaneous T Cell Lymphoma; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BITR2101 (Experimental)
  Interventions: Biological: BITR2101

INTERVENTIONS:
Biological: BITR2101 — TNFR2 monoclonal antibody

SUMMARY:
The goal of this trial is to learn if a new drug, BITR2101, works to treat non-Hodgkin lymphoma (NHL) in adults, with CTCL patients being sought in particular. The trial also seeks to learn about the safety of this drug. This drug is a protein called an antibody. The drug prevents a molecule called a receptor, named TNFR2, from being made. TNFR2 regulates the immune system and provides important signals to lymphoma cells to grow, make more of themselves and survive. When the drug prevents TNFR2 from being produced in lymphoma cells from CTCL patients, those cells died in the laboratory. Therefore, the trial seeks to enroll CTCL patients in particular, in addition to other subtypes of NHL. When the drug prevents the receptor from being made in certain immune cells, there is increased immune activity. Thus, the trial will test if this drug is a new immune therapy that helps the immune system to keep lymphoma under control. In particular, we want to find out if the amount of lymphoma in the body decreases while taking the drug. Patients with autoimmune diseases are not permitted because of this potential increase in immunity brought on by this drug. Patients should have NHL that has been previously treated, that is getting worse on their current therapy, and their doctors think a new treatment is needed. All patients will receive BITR2101 by a 3 hour infusion into a vein, periodically, initially every 3 weeks. There is no placebo in this trial. Visits to the clinic facility will be required, initially at least every week and later less frequently. Patients will be expected to report changes in their health to the clinic staff including new findings and any change in the status of their lymphoma they may be aware of. Patients can continue to receive BITR2101 for up to a year or until their lymphoma worsens. For patients who are clearly benefiting, they may be able to receive BITR2101 for another year.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed relapsed or refractory B cell NHL (DLBCL, MCL, MZL), PTCL or CTCL (MF or SS subtype) as per 2017 World Health Organization classification after at least 2 prior lines of systemic therapy and have received, or are not eligible for, approved or available treatments expected to provide benefit. CTCL patients should be Stage ≥1B through 4 and Stage 1A (see Appendix 1) with plaque disease without treatment options, in which case the patient should be discussed with the sponsor after submitting documentation of disease stage and treatment history. Patients with indolent lymphoid malignancies (CTCL, MZL) must need new treatment regimen in the opinion of the treating Investigator.
* Age ≥18 years.
* Life expectancy ≥3 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Key Exclusion Criteria:

* Patients with prior exposure (up to 12 months) to PD-1/PD-L1 therapies.
* Known hypersensitivity to any excipients that are used in the BITR2101 formulation as noted in Investigator Brochure.
* Autoimmune diseases that have been sufficiently active to require medications in the 3 months before screening, except autoimmune endocrinopathies, such as hypothyroidism, that are stable with hormone-replacement therapy. Including inflammatory diseases such as arthritis, colitis, liver fibrosis, cirrhosis, interstitial fibrosis or chronic obstructive pulmonary disease (COPD). The SRC may allow patients with well controlled arthritis or COPD in the expansion cohort if there is no indication of inflammatory disease flare and no blood cytokine evidence of a systemic inflammatory response in the 3 months prior to enrollment.
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with participating in the protocol.
* History or evidence of clinically significant cardiovascular disease.
* Severe dyspnea, pulmonary dysfunction, or need for continuous supportive oxygen inhalation.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study for the duration of this study or the FU period of an interventional study.
* Prior or current anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy within 4 weeks of the first BITR2101 administration.
* Continuous corticosteroid use exceeding 10 mg/day prednisone or equivalent.

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
to assess the safety and tolerability of BITR2101 administered intravenously every 3 weeks in order to determine the MTD, if any, and to inform the RDE | From enrollment to end of treatment, up to 2 years